CLINICAL TRIAL: NCT03032900
Title: Right Ventricular Dysfunction Incidence After Major Lung Resection, a Prospective Study.
Brief Title: Right Ventricular Dysfunction Incidence After Major Lung Resection
Acronym: RESECHO
Status: Terminated | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF9740
Record Dates: First submitted 2017-01-16; First posted 2017-01-26 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Major Lung Resection; Right Ventricular Dysfunction
Keywords: Major lung resection; Right Ventricular Dysfunction; 2D Strain
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to describe incidence of right ventricular dysfunction after major lung resection with echocardiography criteria.

DETAILED DESCRIPTION:
Few clinical trial studied the incidence of right ventricular dysfunction after major lung resection and time frame of occurrence.

In this prospective observational study the right ventricular function will be mesure with echocardiographic criteria. Echocardiographic exam will be standardised and be realised day before surgery (at the same time that inclusion), day 1, day 2 and day 3 after surgery.

In order to assess prognostic value of right dysfunction after lung resection, data as hospitalization stay, complications and survival will be collected at 6 months.

Cardiac cycles will be recorded and be analysed by a single observer blind to the clinical finding and other echocardiographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Patient older than 18 years
* Major lung surgery (pneumonectomy, lobectomy)

Exclusion Criteria:

* Pre-existing pulmonary arteria hypertension
* Post-operative surgical complication on day 1 to 3 (bleeding, revision surgery)
* Technical difficulty preventing adequate echocardiographic assessment
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major lung surgery
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Right ventricular dysfunction | 5 days
  Without pre-existing pulmonary arteria hypertension, it will be assess with echocardiography criteria : PAPS > 35mmHg or right ventricular dilatation or right systolic markers abnormalities.

SECONDARY OUTCOMES:
Risk factors | 5 days
  Determining risk factors for developing right ventricular failure after pulmonary resection
Time frame to right ventricular dysfunction | 5 days
  Time frame to right ventricular dysfunction
Assessment of 2D strain for right ventricular dysfunctio | 5 days
  Assessment of 2D strain for right ventricular dysfunction
Estimate impact of right ventricular dysfunction on patient prognosis. | 5 days
  Estimate impact of right ventricular dysfunction on patient prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC